CLINICAL TRIAL: NCT05782036
Title: Development, Validation and Clinical Application of a Recovery Scale After Cardiac Surgery: the Fuwai-CRS (Fuwai- Cardiac Recovery Scale)
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-1882
Record Dates: First submitted 2023-02-17; First posted 2023-03-23 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Recovery; Cardiac Surgery; PROM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Item generation
- Cohort 2: Item finalization and validation
- Cohort 3: Clinical application

SUMMARY:
Improving patient recovery after cardiac surgery is a critical priority. While improved surgical techniques have substantially reduced procedural mortality over the past decades, the inherent physiological insult of median sternotomy, cardiopulmonary bypass, and myocardial manipulation continues to impose significant challenges in patient's recovery experience, such as pain, sleep disorders. Paradoxically, this critical recovery phase remains underexplored, as traditional outcome metrics predominantly focus on mortality and major morbidity endpoints. However, no cardiac surgery-specific tools currently exist to adequately capture postoperative recovery experience, creating barriers to optimal care. Accordingly, the investigators aim to develop and validate a recovery scale after cardiac surgery and evaluate its clinical performance compared to the generic scale (QoR-15)

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery

Exclusion Criteria:

* Emergency surgery
* Age ≤ 18 years
* Refuse to participate in this study
* prolonged postoperative mechanical ventilation exceeding 24 hours reoperation or perioperative death

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient aged 18 years or older, undergoing elective cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 3043 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Death or unplanned readmission | 3-month post operative

SECONDARY OUTCOMES:
In-hospital mortality | From surgery to discharge, up to 7 days
  Occurrence of death during hospitalization
In-hospital stroke | From surgery to discharge, up to 7 days
  Occurrence of stroke during hospitalization
In-hospital myocardial infarction | From surgery to discharge, up to 7 days
  Occurrence of myocardial infarction during hospitalization
In-hospital acute renal failure | From surgery to discharge, up to 7 days
  Occurrence of acute renal failure during hospitalization
In-hospital sternal wound infection | From surgery to discharge, up to 7 days
  Occurrence of sternal wound infection during hospitalization
In-hospital reoperation | From surgery to discharge, up to 7 days
  Occurrence of reoperation during hospitalization
Length of hospital stay | Approximately 7 days
  Length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China